CLINICAL TRIAL: NCT07244250
Title: Result of Root Canal Treatment in General Dentistry
Brief Title: The Present Study Aims to Follow up on All Root Canal Treatments Performed During the Year 2023 Within the Public Dental Services of the Counties of Jönköping, Kalmar, and Östergötland, Sweden. The Study is Entirely Observational in Nature.
Status: Not yet recruiting | Type: Observational
Sponsor: Region Jönköping County (Other Government)
Collaborators: Region Östergötland (Other); Kalmar County Council (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-04871-02
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Endodontic Treatment; Apical Periodontitis; Quality
Keywords: Root canal treatment; Apical periodontitis; Root filling
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients who have received root canal treatment in the Public Dental Service in the counties of Jönköping, Kalmar and Östergötland

SUMMARY:
Each year, nearly 200,000 teeth undergo root canal treatment in Sweden, most of them within general dental care. However, studies that evaluate the outcomes of root canal treatments have almost exclusively been conducted at specialist or university clinics, where treatment conditions differ from everyday practice in general dentistry. Moreover, the design of such studies often limits the ability to generalize their findings to routine clinical settings.

These earlier studies suggest that root canal treatment is a predictable procedure-about 80-90% of treated teeth become free from infection, 90% of patients experience no pain, and approximately 90% of root-filled teeth remain in the mouth six years after treatment. Still, the results from these studies cannot easily be applied to general dental care. This has been confirmed by large-scale epidemiological studies using X-rays to assess the technical quality of performed root fillings and to detect signs of disease. These studies have shown that many root fillings exhibit technical shortcomings, and a significant proportion of root-treated teeth have persistent infections.

The current study aims to increase understanding of the factors that may explain why the results of root canal treatment in general dental practice appear to differ from those in specialist care. Based on epidemiological data, it is estimated that about 35% of teeth treated with root canal therapy in general dental practice still show signs of disease after treatment. What happens to these patients is largely unknown. Evidence suggests that teeth with persistent apical periodontitis rarely cause discomfort, and the condition often goes unnoticed.

In the first part of the study, only patients who have already received treatment will be invited to participate, making this a retrospective study. Because it takes several years to evaluate the outcome of a root canal treatment, all patients aged 20 years and older who had a tooth root-filled in 2023 within the Public Dental Services of Jönköping, Kalmar, or Östergötland counties will be offered a free clinical and radiological examination-thus a three-year follow-up. The examination is entirely painless.

In the second part of the study, patients with a root-filled tooth showing persistent disease will be offered a five-year follow-up (2026-2031). They will be grouped according to whether they choose to have further treatment or leave the condition untreated. This second phase will therefore constitute a prospective follow-up.

ELIGIBILITY:
Inclusion Criteria:

• All patients who have received and completed a root canal treatment in the Public Dental Service in the counties of Jönköping, Kalmar and Östergötland in 2023.

Exclusion Criteria:

• All patients who decline participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received and completed a root canal treatment in the Public Dental Service in the counties of Jönköping, Kalmar and Östergötland in 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Posttreatment frequency of apical periodontitis | three year follow-up
  Apical periodontitis as defined as a periapcal radiolucency on an intra oral radiograph
Posttreatment frequency of apical periodontitis | From completion of treatment to three year follow-up
  Apical periodontitis as defined as a periapical radiolucency

IPD SHARING:
Plan to Share IPD: Undecided